CLINICAL TRIAL: NCT02806505
Title: A Randomized, Open-Label, Multicenter, Parallel Group Study Evaluating the Efficacy and Safety of 135 μg and 90 μg of PEGASYS® Given as Monotherapy to Patients With Chronic Hepatitis C and End-Stage Renal Disease Undergoing Hemodialysis
Brief Title: HELPS Study - A Study of Peginterferon Alfa-2a (Pegasys) in Patients With Chronic Hepatitis C (CHC) and End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MV17149
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- Peginterferon alfa-2a 135 microgram (mcg) (Experimental): Chronic Hepatitis C participants with end-stage renal disease undergoing hemodialysis will receive Peginterferon alfa-2a 135 mcg subcutaneously (SC) once weekly up to Week 48.
  Interventions: Drug: Peginterferon alfa-2a
- Peginterferon alfa-2a 90 mcg (Experimental): Chronic Hepatitis C participants with end-stage renal disease undergoing hemodialysis will receive Peginterferon alfa-2a 90 mcg SC once weekly up to Week 48.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Chronic Hepatitis C participants with end-stage renal disease undergoing hemodialysis will receive Peginterferon alfa-2a either 135 or 90 mcg SC once weekly up to Week 48.
  Other Names: Pegasys

SUMMARY:
This study evaluated the safety and efficacy of peginterferon alfa-2a monotherapy in participants with Chronic Hepatitis C (CHC) who have End-Stage Renal Disease (ESRD) and were undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Serum hepatitis C virus ribonucleic acid (HCV RNA) quantifiable at greater than (>) 600 IU/mL
* Liver biopsy consistent with chronic hepatitis C infection obtained within 2 years of enrollment
* Compensated liver disease without cirrhosis
* Participants with end-stage renal disease undergoing hemodialysis
* Negative serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile participants must have been using effective contraception during treatment with study drug

Exclusion Criteria:

* Interferon therapy at any previous time
* Liver cirrhosis
* Signs and symptoms of hepatocellular carcinoma
* History or other evidence of decompensated liver disease
* Any investigational drug less than or equal to 6 weeks prior to the first dose of study drug
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Poorly controlled diabetes
* Thyroid dysfunction not adequately controlled
* Evidence of severe retinopathy or clinically relevant ophthalmological disorder
* Severe hyperparathyroidism defined as intact Parathyroid Hormone (PTH) > 800 picogram/milliliter (pg/mL)
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment ≤ 6 months prior to the first dose of study drug
* Acute renal failure
* Women with ongoing pregnancy or breast feeding
* Positive test at screening for anti-HAV IgM Ab (hepatitis A virus immunoglobulin M antibody), hepatitis B surface antigen (HBsAg), anti-HBc (hepatitis B core) IgM Ab, anti-HIV (human immunodeficiency virus) Ab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (20):
- Austria (2):
  - Graz
  - Vienna
- Brazil (5):
  - Brasília
  - Porto Alegre
  - Sao Jose Rio Preto
  - São Luís
  - São Paulo
- France (6):
  - Créteil
  - Le Kremlin-Bicêtre
  - Marseille
  - Paris
  - Strasbourg
  - Toulouse
- Greece (2):
  - Athens
  - Nikaia
- Medan, Indonesia
- Cagliari, Italy
- Turkey (Türkiye) (2):
  - Istanbul
  - Izmir
- Abu Dhabi, United Arab Emirates

REFERENCES:
- [Derived] Prabhu AR, Rao IR, Nagaraju SP, Rajwar E, Venkatesh BT, Nair N S, Pai G, Reddy NP, Suvarna D. Interventions for dialysis patients with hepatitis C virus (HCV) infection. Cochrane Database Syst Rev. 2023 Apr 25;4(4):CD007003. doi: 10.1002/14651858.CD007003.pub3. PMID 37096802

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 85 participants were randomly assigned to the two treatment groups (Peginterferon alfa-2a 135 mcg/week and Peginterferon alfa-2a 90 mcg/week). A total of 4 randomized participants did not receive any study drug.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg
Started | 38 | 43
Completed | 28 | 32
Not Completed | 10 | 11
Not completed — Adverse event/intercurrent illness | 1 | 3
Not completed — Death | 4 | 0
Not completed — Did not cooperate/refused treatment | 3 | 3
Not completed — Failure to return | 0 | 1
Not completed — Insufficient therapeutic response | 2 | 4

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis population included all the randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg | Total
Number analyzed (Participants) | 38 | 43 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.26) | 42.9 (11.26) | 43.5 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 23 | 34 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response (SVR) at 24 Weeks After End of Treatment
Description: SVR was defined as the percentage of patients with undetectable HCV RNA. SVR rate was calculated as the number of participants with an undetectable HCV RNA divided by the number of participants of the respective participant population. The last single HCV RNA less than (<) 50 international units per millilitre (IU/mL) measured >=140 days after treatment end (i.e., >= 20 weeks after treatment end) was used to determine SVR. Participants without measurements in this time window were considered to be nonresponders.
Time Frame: 24 weeks after end of treatment (Week 72)
Population: The ITT analysis population included all the randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg
Number analyzed (Participants) | 38 | 43
percentage of participants | 39.5 [24.0 to 56.6] | 34.9 [21.0 to 50.9]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a 135 Microgram (mcg) vs Peginterferon Alfa-2a 90 mcg; The odds ratio is the ratio of the odds of a response in the Peginterferon alfa-2a 135 mcg group with the odds of a response in the Peginterferon alfa-2a 90 mcg group; Test type: Superiority or Other; p = 0.6746, Cochran-Mantel-Haenszel — Assessed by Cochran-Mantel-Haenszel test stratified by country (Brazil, France, Other) and HCV genotype (1 vs. non-1); Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.49 to 3.06]

2. Secondary Outcome: Percentage of Participants With Virological Response (Non-detectable Hepatitis C Virus-ribonucleic Acid [HCV RNA]) at End of Treatment (EOT)
Description: Virological response at the end of study treatment was defined as the percentage of participants with undetectable HCV RNA. This response rate at end of treatment was calculated as the number of participants with undetectable HCV RNA divided by the number of participants of the respective participant population.
Time Frame: EOT (Week 48)
Population: The ITT analysis population included all the randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg
Number analyzed (Participants) | 38 | 43
percentage of participants | 57.9 [40.8 to 73.7] | 48.8 [33.3 to 64.5]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a 135 Microgram (mcg) vs Peginterferon Alfa-2a 90 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3923, Cochran-Mantel-Haenszel — Assessed by Cochran-Mantel-Haenszel test stratified by country (Brazil, France, Other) and HCV genotype (1 vs. non-1); Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.60 to 3.76]

3. Secondary Outcome: Percentage of Participants With Virological Response (at Least a 2-log 10 Decrease in HCV RNA as Compared With Baseline or Unquantifiable [Less Than {<} 600 International Unit/Milliliter {IU/mL}] or Undetectable HCV RNA [< 50 IU/mL]) at Week 12 and 24
Description: Virological response at Weeks 12 and 24 was computed as the percentage of participants with at least a 2-log 10 decrease in HCV RNA at Weeks 12 and 24 as compared with baseline or with an unquantifiable (< 600 IU/mL) or an undetectable HCV RNA test result (< 50 IU/mL) at Week 12 and at Week 24, calculated as the number of participants meeting this criterion divided by the number of participants of the respective participant population.
Time Frame: Weeks 12 and 24
Population: The ITT analysis population included all the randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg
Number analyzed (Participants) | 38 | 43
percentage of participants
  Week 12 | 71.1 [54.1 to 84.6] | 69.8 [53.9 to 82.8]
  Week 24 | 65.8 [48.6 to 80.4] | 72.1 [56.3 to 84.7]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a 135 Microgram (mcg) vs Peginterferon Alfa-2a 90 mcg; Week 12: The odds ratio is the ratio of the odds of a response in the Peginterferon alfa-2a 135 mcg group with the odds of a response in the Peginterferon alfa-2a 90 mcg group; Test type: Superiority or Other; p = 0.8843, Cochran-Mantel-Haenszel — Assessed by Cochran-Mantel-Haenszel test stratified by country (Brazil, France, Other) and HCV genotype (1 vs. non-1); Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.43 to 2.68]
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a 135 Microgram (mcg) vs Peginterferon Alfa-2a 90 mcg; Week 24: The odds ratio is the ratio of the odds of a response in the Peginterferon alfa-2a 135 mcg group with the odds of a response in the Peginterferon alfa-2a 90 mcg group; Test type: Superiority or Other; p = 0.5866, Cochran-Mantel-Haenszel — Assessed by Cochran-Mantel-Haenszel test stratified by country (Brazil, France, Other) and HCV genotype (1 vs. non-1); Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.28 to 2.04]

ADVERSE EVENTS:
Time Frame: Baseline up to follow up period (Week 72)
Description: An adverse event was defined as any untoward medical occurrence that occurred during the course of the trial after study treatment had started.
Arm/Group | Peginterferon Alfa-2a 135 Microgram (mcg) | Peginterferon Alfa-2a 90 mcg
Serious Adverse Events (participants affected / at risk) | 14/38 | 14/43
Other Adverse Events (participants affected / at risk) | 30/38 | 38/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 135 Microgram (mcg) (N=38) | Peginterferon Alfa-2a 90 mcg (N=43)
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Hypertrophic cardiomyopathy (Cardiac disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Gene mutation (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1
Medical observation (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ventricle rupture (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a 135 Microgram (mcg) (N=38) | Peginterferon Alfa-2a 90 mcg (N=43)
Anaemia (Blood and lymphatic system disorders) | 14 | 14
Hyperparathyroidism secondary (Endocrine disorders) | 4 | 6
Hypothyroidism (Endocrine disorders) | 4 | 0
Conjunctivitis (Eye disorders) | 1 | 3
Eye pain (Eye disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 7 | 7
Chills (General disorders) | 3 | 0
Fatigue (General disorders) | 6 | 7
Influenza like illness (General disorders) | 6 | 6
Malaise (General disorders) | 2 | 1
Pyrexia (General disorders) | 5 | 7
Oral herpes (Infections and infestations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 9 | 13
Depression (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 5 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.